CLINICAL TRIAL: NCT02151838
Title: The Thai Red Cross AIDS Research Centre
Brief Title: The Thai Red Cross Society Prevention of Mother-To-Child Transmission of HIV (TRCS PMTCT) Program
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: TRCS PMTCT
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: HIV-infected Pregnant Women Who Request HAART From the TRCSPMTCT
Keywords: HIV-infected pregnant women who request HAART from the TRCSPMTCT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess the safety and the efficacy of Highly Active Anti-Retroviral Treatment (HAART) for the Prevention of Mother-To-Child Transmission of HIV (PMTCT)

DETAILED DESCRIPTION:
1. To describe characteristics of HIV-infected pregnant women who request HAART from the Thai Red Cross Society PMTCT (TRCS PMTCT) program
2. To study adverse pregnancy outcomes among HIV-infected pregnant women who receive HAART
3. To study adverse events in infants born to women who receive HAART during pregnancy
4. To evaluate risk factors for HAART-related toxicities and for perinatal HIV transmission
5. To establish the pilot model of care for HIV-infected pregnant women in middle income country

ELIGIBILITY:
Inclusion Criteria:

Volunteers meeting all of the following criteria will be considered eligible for enrollment in the study:

1. HIV-infected pregnant women (as defined by the hospital)
2. Choose to start HAART according to protocol and do not want to receive antiretroviral treatment provided by the other health care systems
3. Understand the study and sign informed consent form. Persons who cannot read will have the consent form read to them by a study staff and they can give informed consent by using thumb print.
4. Availability for follow-up for the planned study duration

Exclusion Criteria:

Volunteers meeting any of the following criteria will be excluded from the study:

1.Persons who have a history of a medical or psychiatric disorder by interview and physical examination according to standard practices, that in the judgment of the treating physician, would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent.

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population will be HIV-infected pregnant women who request HAART from the TRCS PMTCT program. These pregnant women will be under the care of the health care teams in 30 hospitals throughout Thailand which have registered with the TRCS PMTCT program since April 2004
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
HIV-infected pregnant women | 18 months
  Choose to start HAART according to protocol and do not want to receive antiretroviral treatment provided by the other health care systems

CONTACTS AND LOCATIONS:
Locations (1):
- The Thai Red Cross AIDS Research Centre, Pathum Wan, Bangkok, Thailand